CLINICAL TRIAL: NCT01196052
Title: A Multicenter, Multinational Phase II Study to Assess the Clinical Safety and Feasibility of Trastuzumab Emtansine Sequentially With Anthracycline-based Chemotherapy, as Adjuvant or Neoadjuvant Therapy for Patients With Early Stage HER2-positive Breast Cancer
Brief Title: A Study of Trastuzumab Emtansine (T-DM1) Sequentially With Anthracycline-based Chemotherapy, as Adjuvant or Neoadjuvant Therapy for Patients With Early Stage Herceptin (HER)2-positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO22857; TDM4874g (Other: Genentech, Inc.)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (1):
- Trastuzumab emtansine (Experimental): Trastuzumab emtansine 3.6 mg/kg was administered intravenously on Day 1 of each 3-week treatment cycle up to a maximum of 17 cycles.
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine — Trastuzumab emtansine was provided as a single-use lyophilized formulation in a glass vial.
  Other Names: T-DM1

SUMMARY:
This single-arm open-label study assessed the safety, feasibility, and efficacy of trastuzumab emtansine (T-DM1) after the completion of anthracycline-based adjuvant/neoadjuvant chemotherapy in patients with early HER2-positive breast cancer. Patients received T-DM1 3.6 mg/kg intravenously on Day 1 of each 3-week cycle, for up to 17 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Locally advanced, inflammatory, or early stage, unilateral, and histologically confirmed invasive breast cancer documented at a local laboratory (patients with inflammatory breast cancer must be able to have a core needle biopsy).
* Herceptin (HER)2-positive tumor, confirmed by central testing using immunohistochemistry (IHC) and in situ hybridization (ISH) methods.
* Willingness to receive anthracycline-based chemotherapy or have received doxorubicin/cyclophosphamide (AC) OR 5-fluorouracil (FU)/epirubicin/ cyclophosphamide (FEC) in a similar dose and schedule as described in the protocol as part of neoadjuvant or adjuvant treatment.
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective, non-hormonal form of contraception or 2 effective forms of non-hormonal contraception by the patient and/or partner. Contraception use must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment. Male patients should use condoms for the duration of the study. Specific country requirements will be followed.
* Negative results of serum pregnancy test for premenopausal women of reproductive capacity and for women < 12 months after menopause.
* Patients may enroll before or after AC/FEC chemotherapy has completed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, biochemistry, and cardiac assessments.

Exclusion Criteria:

* Stage IV breast cancer or bilateral breast cancer.
* Pregnant or breastfeeding women.
* History of other malignancy within the previous 5 years, except contralateral breast cancer and ductal carcinoma in situ (DCIS)/lobular carcinoma in situ (LCIS), appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with outcome similar to those mentioned above.
* Radiation therapy, immunotherapy, or biotherapy within 5 years before study enrollment; non-cardiotoxic chemotherapy for malignancy treated > 5 years before study enrollment is allowed. Patients receiving AC/FEC in a similar fashion to the study treatment prescribed for adjuvant or neoadjuvant treatment of breast cancer will be allowed to enroll in the study after the completion of their AC/FEC. No other prior history of cardiotoxic chemotherapy is allowed.
* Active cardiac history.
* Current chronic daily treatment with oral corticosteroids or equivalent.
* Patients with severe dyspnea at rest or requiring supplementary oxygen therapy.
* Active, unresolved infections at screening.
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
* Major surgery within 4 weeks before enrollment that is unrelated to the breast cancer.
* Patients for whom concomitant radiotherapy + T-DM1 may be contraindicated yet radiation therapy is planned.
* Known hypersensitivity to any of the study drugs or derivatives, including murine proteins.
* Grade ≥ 2 peripheral neuropathy at Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (14):
  - Fort Myers, Florida
  - Lafayette, Indiana
  - Scarborough, Maine
  - Kensignton, Maryland
  - Boston, Massachusetts
  - Springfield, Missouri
  - Omaha, Nebraska
  - Lake Success, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Sioux Falls, South Dakota
  - Nashville, Tennessee
  - San Antonio, Texas
  - Tacoma, Washington
- Belgium (2):
  - Brussels
  - Wilrijk
- France (3):
  - Besançon
  - Montpellier
  - Saint-Herblain
- Germany (6):
  - Bielefeld
  - Cologne
  - Frankfurt am Main
  - Hamburg
  - Mönchengladbach
  - Rostock
- Italy (7):
  - San Giovanni Rotondo, Apulia
  - Bologna, Emilia-Romagna
  - Lecco, Lombardy
  - Milan, Lombardy
  - Candiolo, Piedmont
  - Perugia, Umbria
  - Vicenza, Veneto
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Tula
- Seoul, South Korea
- Spain (4):
  - Barcelona, Barcelona
  - Jaén, Jaen
  - Lleida, Lerida
  - Madrid, Madrid

REFERENCES:
- [Derived] Krop IE, Suter TM, Dang CT, Dirix L, Romieu G, Zamagni C, Citron ML, Campone M, Xu N, Smitt M, Gianni L. Feasibility and cardiac safety of trastuzumab emtansine after anthracycline-based chemotherapy as (neo)adjuvant therapy for human epidermal growth factor receptor 2-positive early-stage breast cancer. J Clin Oncol. 2015 Apr 1;33(10):1136-42. doi: 10.1200/JCO.2014.58.7782. Epub 2015 Feb 23. PMID 25713436

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab Emtansine
Started | 153
Received Trastuzumab Emtansine | 148
Completed | 130
Not Completed | 23
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 1
Not completed — Noncompliance to Protocol Requirements | 2
Not completed — Reason not Specified | 5
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Enrolled participant population: All participants enrolled in the study.
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Cardiac Event Within 12 Weeks After the Start of Trastuzumab Emtansine Treatment
Description: A cardiac event was defined as death from a cardiac cause or severe congestive failure (New York Heart Association [NYHA] Class III or IV) with a decrease in left ventricular ejection fraction (LVEF) of ≥ 10% from Baseline to an LVEF of < 50%.
Time Frame: Baseline to 12 weeks after the start of trastuzumab emtansine treatment
Population: Cardiac-safety evaluable population: All participants who received at least 1 dose of T-DM1 and met either of the following 2 criteria: (1) Had an echocardiogram/multiple-gated acquisition assessment by 12 weeks after the first dose of T-DM1 or (2) discontinued study treatment because of cardiac toxicity prior to completion of 4 cycles of T-DM1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 143
Percentage of participants | 0 [0.00 to 2.45]

2. Primary Outcome: Adverse Events, LVEF Function, and Deaths
Description: The following percentages of participants are reported: At least 1 adverse event while receiving T-DM1; at least 1 serious adverse event while receiving T-DM1; an adverse event leading to discontinuation, dose delay, or dose reduction of trastuzumab emtansine treatment; symptomatic cardiac dysfunction; and asymptomatic decline in left ventricular ejection fraction (LVEF). An asymptomatic LVEF decline was defined as a LVEF < 50% and a maximum decrease ≥ 10% from Baseline. The percentage of participants who died is reported.
Time Frame: From the start to the end of trastuzumab emtansine treatment (up to 51 weeks)
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 148
Percentage of participants
  At least 1 adverse event (AE) | 98.6
  At least 1 serious adverse event | 10.1
  An AE leading to treatment discontinuation | 13.5
  An AE leading to dose delay | 29.1
  An AE leading to dose reduction | 21.6
  Symptomatic cardiac dysfunction | 0.0
  An asymptomatic decline in LVEF | 2.7
  Deaths | 0

3. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event During Concurrent Radiotherapy With Trastuzumab Emtansine Treatment
Time Frame: From the start to the end of concurrent radiotherapy (up to 51 weeks)
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine. Only participants who received concurrent radiotherapy were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 39
Percentage of participants | 94.9

4. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event During Concurrent Hormonal Therapy With Trastuzumab Emtansine Treatment
Time Frame: From the start to the end of concurrent hormonal therapy (up to 51 weeks)
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine. Only participants who received concurrent hormonal therapy were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 62
Percentage of participants | 69.4

5. Secondary Outcome: Percentage of Participants Who Completed the Planned Duration of Trastuzumab Emtansine Treatment
Description: Participants were to receive up to a total of 17 cycles of trastuzumab emtansine. If trastuzumab was given concurrently with either the optional docetaxel or optional radiation, then the number of 3-week cycles of trastuzumab therapy was subtracted from the planned 17 cycles of trastuzumab emtansine therapy.
Time Frame: From the start to the end of trastuzumab emtansine treatment (up to 51 weeks)
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 148
Percentage of participants | 82.4

6. Secondary Outcome: Percentage of Participants Who Completed ≥ 95% of the Planned Radiotherapy Treatment With Concurrent Trastuzumab Emtansine Administration Without Significant (> 5 Days) Delay
Time Frame: From the start to the end of radiotherapy treatment (up to 51 weeks)
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine. Only participants who received concurrent radiotherapy and who had radiotherapy dose information reported were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 38
Percentage of participants | 94.7

7. Secondary Outcome: Percentage of Participants With a Pathological Complete Response
Description: Pathological complete response was defined as the absence of invasive neoplastic cells at microscopic examination of the primary tumor and lymph nodes after surgery following primary systemic therapy. Pathological complete response was evaluated in participants treated with neoadjuvant therapy doxorubicin/cyclophosphamide-5-fluorouracil/epirubicin/cyclophosphamide followed by 1 or more doses of trastuzumab emtansine and who underwent surgery.
Time Frame: Day of surgery
Population: Efficacy analysis population: All participants who enrolled in the neoadjuvant setting and received surgery, after completing 4 cycles of trastuzumab emtansine treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 50
Percentage of participants | 56.0 [41.3 to 69.6]

8. Secondary Outcome: Disease-free Survival at Month 12
Description: Disease-free survival was defined as the time from date of first protocol treatment for adjuvant patients or date of surgery for neoadjuvant patients to disease recurrence, occurrence of invasive contralateral breast cancer, other second primary cancer (excluding non-breast second primary), or death, whichever occurred first.
Time Frame: From the start of trastuzumab emtansine for adjuvant patients and from the date of surgery for neoadjuvant patients to 12 months later
Population: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine.
  Due to too few events, the analysis of disease-free survival was not performed.
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Safety-evaluable population: All participants who received at least 1 dose of trastuzumab emtansine.
  All adverse events that occurred while participants were receiving trastuzumab emtansine are reported.
Arm/Group | Trastuzumab Emtansine
Serious Adverse Events (participants affected / at risk) | 15/148
Other Adverse Events (participants affected / at risk) | 146/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine (N=148)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=148)
Asthenia (General disorders) | 45
Fatigue (General disorders) | 34
Pyrexia (General disorders) | 39
Mucosal Inflammation (General disorders) | 10
Influenza Like Illness (General disorders) | 20
Chills (General disorders) | 19
Oedema Peripheral (General disorders) | 9
Nausea (Gastrointestinal disorders) | 56
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 25
Dry Mouth (Gastrointestinal disorders) | 20
Stomatitis (Gastrointestinal disorders) | 9
Abdominal Pain Upper (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 12
Abdominal Pain (Gastrointestinal disorders) | 14
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 8
Gingival Bleeding (Gastrointestinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 24
Pruritus (Skin and subcutaneous tissue disorders) | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 9
Nail Disorder (Skin and subcutaneous tissue disorders) | 9
Headache (Nervous system disorders) | 55
Dysgeusia (Nervous system disorders) | 13
Neuropathy Peripheral (Nervous system disorders) | 18
Peripheral Sensory Neuropathy (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 16
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 16
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9
Nasopharyngitis (Infections and infestations) | 20
Upper Respiratory Tract Infection (Infections and infestations) | 15
Urinary Tract Infection (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 32
Anaemia (Blood and lymphatic system disorders) | 13
Radiation Skin Injury (Injury, poisoning and procedural complications) | 12
Aspartate Aminotransferase Increased (Investigations) | 19
Alanine Aminotransferase Increased (Investigations) | 18
Conjunctivitis (Eye disorders) | 9
Dry Eye (Eye disorders) | 8
Decreased Appetite (Metabolism and nutrition disorders) | 18
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hot Flush (Vascular disorders) | 20
Hypertension (Vascular disorders) | 8
Insomnia (Psychiatric disorders) | 12
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 11
Breast Pain (Reproductive system and breast disorders) | 10
Vertigo (Ear and labyrinth disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.